CLINICAL TRIAL: NCT01051895
Title: Randomized Controlled Trial Comparing Routine Colposcopy to HPV Testing to Identify Persistent or Recurrent High Grade Cervical Cancer Precursors
Brief Title: Colposcopy Versus HPV Testing to Identify Persistent Cervical Precancers
Acronym: CoHIPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Terry Fox Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09.078
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: High Grade Cervical Intra-epithelial Neoplasia
Keywords: Cervical intra-epithelial neoplasia; Colposcopy; HPV DNA testing; treatment failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV testing (Experimental): Women randomized to this arm will undergo high risk HPV DNA testing using Hybrid Capture 2®.
  Interventions: Other: high risk HPV DNA testing
- Routine colposcopy (Active Comparator): Women will be followed in the colposcopy clinic as usual, with no standardized protocol, tests are left at the discretion of the treating physician, in order to document routine proactive. We will document all procedures (biopsies, endocervical curettage, cytology, etc) and their outcome.
  Interventions: Other: Active comparator: Routine colposcopy

INTERVENTIONS:
Other: high risk HPV DNA testing — Specimens will be collected with a cervical cytobrush and cervical cells will be resuspended in 2 ml of Preservcyt® (Hologic LP), a liquid cytology preservation media. 75µl of processed sample will be hybridized with 25 µl of probe B mixture. The assay is completed as a standard enzyme immunoassay with the addition of a dioxetane-based chemiluminescent substrate. Specimens will be considered positive for HPV if the ratio of RLUs of the specimen to the mean RLUs of triplicates of positive control (at 1 pg per ml or 5000 copies of HPV genome per test) is at least one.
  Other Names: Hybrid Capture 2®
  Arms: HPV testing
Other: Active comparator: Routine colposcopy — Women will undergo colposcopy, with no standardized protocol; tests are left at the discretion of the treating physician, in order to document routine proactive. We will document all procedures (biopsies, endocervical curettage, cytology, etc) and their outcome.
  Arms: Routine colposcopy

SUMMARY:
This trial will compare HPV testing to the routine colposcopy in the follow-up of women treated for cervical high grade lesions. Women will be assigned randomly (by chance) after treatment of cervical pre-cancer to be either (1) followed-up by colposcopy, or (2) undergo HPV testing. Women found to have disease by either strategy will be offered re-treatment. For the next 2 years participants will undergo yearly, in depth, evaluation to assess the cervix for precancer. We will then be able to compare which of the 2 follow-up strategies worked best.

DETAILED DESCRIPTION:
Background and rational: Cervical cancer ranks twelfth in terms of cancer mortality in Canadian women, but remains the second most frequent cancer in Canadian women aged 20-44. Fortunately, its natural history makes it an ideal candidate for successful prevention. Cervical cancer and its precursors are caused by a persistent infection of the cervical epithelium by one of the 15 oncogenic (or high risk) types of human papillomaviruses (HPVs). The preinvasive changes of cervical intra-epithelial neoplasia (CIN) can be identified through cervical cytology (also known as the Pap test). When cellular abnormalities are identified, women are referred for diagnostic testing. High-grade precursor lesions (CIN2/3) carry a high risk of progression to invasive cancer and for this reason their treatment is recommended. Treatment success rates of CIN2/3 are 85%. However, those who fail treatment need to be identified promptly because their risk of invasive disease is increased more then 10 fold. The current strategy used in Canada to identify treatment failures consists of a follow-up every 6 months in colposcopy clinics for 2 years. Recent research underlines the fact that routine colposcopy is unreliable and may miss significant lesions. The identification of oncogenic HPV DNA in the cervical secretions is known as HPV testing. A few studies have investigated the use of HPV testing in the identification of treatment failures. Although they point to a very good sensitivity (90-95%) there were methodological limitations: studies were small; the HPV test used was often not suitable for clinical laboratory use; endpoints were not assessed by histological confirmation. Most importantly, none compared HPV testing to colposcopy, the strategy used in Canada. Research question: Is HPV testing more sensitive than routine colposcopy to identify CIN2/3 treatment failures? Methodology: Design: We propose a parallel randomized controlled trial, where participants will be randomized 1:1 to routine colposcopy vs. HPV testing after treatment of CIN2/3 lesions. Study Population: Women treated for high-grade precursor lesions. Exclusion criteria are: pregnancy, less than 18 years of age, known immunosuppression or immunodeficiency, unable to provide informed consent. Study interventions: (1) HPV testing with Hybrid Capture 2. (2) Routine colposcopy. In order to evaluate the performance of the current follow-up strategy, there will be no standardized protocol for the colposcopy intervention, but documentation of procedures will be done. Patients will receive the study interventions 6 months after treatment. All participants will undergo expert diagnostic assessment at 12 and 24. Sample size calculation and recruitment rate. The sample size was calculated to have 80% power to detect an increase in sensitivity of 15%, with an alpha set at 0.05 (double sided test). Assuming a conservative baseline sensitivity of 70% for colposcopy, 134 cases of recurrent/persistent disease will be necessary in each study group. Assuming a 15% failure rate of treatment and a 20% drop out rate, a total of 2250 participants will need to be accrued. Recruitment will take place in high volume colposcopy clinics across Canada over 2 years. Analysis: The primary analysis will consist of the comparison of the diagnostic indices of the 2 follow-up strategies: sensitivity, specificity, positive and negative predictive values (with their 95% asymptotic confidence intervals). Cumulative persistent/recurrent cases identified during the 2 year follow-up will make up the case group. Since all participants will undergo expert diagnostic assessment. No subgroup analysis will be performed. 4. Expected contribution: The result from this trial will provide high quality data on which to base management recommendation. If HPV testing is found to be more sensitive than routine colposcopy, follow-up of treated lesion may occur mainly in primary care physician's office with HPV testing, reducing costs, and making it possible to focus colposcopy activities on a group of women truly at risk of significant disease.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old 19 in British Columbia, Nova Scotia and Newfoundland)
* Understands English or French (for sites where French speaking coordinator is available)
* Is treated for biopsy proven CIN II, III or AIS
* Understands study procedures, available alternatives treatment, risks related to study, and accepts voluntarily to participate by signing the ICF.

Exclusion Criteria:

* has been treated for cervical cancer or pre-cancer in the past
* Participant has known immunosuppression or immunodeficiency
* Planned hysterectomy
* Participant is receiving or has received one of the following treatment :

  * Immunosuppressive therapy in the three months prior to enrollment
  * Corticosteroid therapy in the two weeks prior to enrollment
  * Two or more courses of corticosteroids (orally or parenterally) lasting at least one week in duration in the year prior to enrollment (inhalation, nasal or topical corticosteroids are permitted)
* There is a strong probability that the participant will not follow the procedures of study, will not come to its appointment, or plans a delocalization throughout study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2253 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of HPV testing and sensitivity of routine colposcopy to identify CIN2 or worse disease after treatment for CIN 2/3 | 6 months post treatment

SECONDARY OUTCOMES:
The area under the respective ROC curves (HPV testing and routine colposcopy) | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Mayrand, MD,PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre de recherche du CHUM, Montreal, Quebec, Canada